CLINICAL TRIAL: NCT04031937
Title: Sensory and Psychomotor Profile in Depression
Acronym: DEPCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, Principal Investigator, Centre Hospitalier Esquirol
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018-A02055-50
Record Dates: First submitted 2019-06-13; First posted 2019-07-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
Keywords: depression; psychomotor assessment; sensory profile; perception; motricity
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- major depressive disorder (Active Comparator): psychometric scales psychomotor assessment
  Interventions: Other: Psychomotor assessment
- Control (Active Comparator): psychometric scales psychomotor assessment
  Interventions: Other: Psychomotor assessment

INTERVENTIONS:
Other: Psychomotor assessment — the intervention include a depression scale, an anxiety scale, a sensory profile scale, a body image questionnaire, a self-esteem questionnaire, a psychomotor retardation scale and a standardized assessment of : muscle tone (dangling and extensibility); gross motor skills (walks, jump, static balance, dynamic balance); manual performance; manual praxis; adaptation of rhythm; manual gnosis; executive function

SUMMARY:
Despite a possible psychomotor retardation during a depressive episode, standardized psychomotor assessment is rare. So, other possible psychomotor disorders or neurological "soft signs" are not known in depression.

The investigator propose in this study to explore the psychomotor characteristics of patients with a major depressive disorder from the realization of a psychomotor assessment in comparison with adult without depressive disorder (control). It will be specifically assess muscle tone, gross motor skills, praxis, body schema and the body image and the perceptions.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder according to the DSM-5
* aged to 18 from 65 years old

Exclusion Criteria:

* psychiatric comorbidity (bipolar, addiction, eating disorder, personality disorder, obsessional compulsive disorder)
* antipsychotic drug
* taken care in psychomotor therapy previously
* electroconvulsive therapy
* medical history of neurologic disease, neurodevelopmental disorder, sensory disability
* Constraint Hospitalization
* under legal protection
* pregnant
* lack of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
% of patients with a distinctive feature at the sensory profile questionnaire from the AASP | At inclusion
  Scores at the AASP psychomotor battery are considered. A failure is considered from a result <1SD compared to the control group.
% of patients with a failure at the muscle tone test from the NP-MOT battery | At inclusion
  Scores at the NP-MOT psychomotor battery are considered. A failure is considered from a result <1SD compared to the control group.
% of patients with a failure at the gross motor test from the NP-MOT battery | At inclusion
  Scores at the NP-MOT psychomotor battery are considered. A failure is considered from a result <1SD compared to the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paquet A, Lacroix A, Calvet B, Girard M. Psychomotor semiology in depression: a standardized clinical psychomotor approach. BMC Psychiatry. 2022 Jul 15;22(1):474. doi: 10.1186/s12888-022-04086-9. PMID 35841086